CLINICAL TRIAL: NCT01443871
Title: Effect of Essential Oils in Aromatherapy on Emotional Relaxation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Phayao (Other)
Responsible Party: Principal Investigator, Surasak Saokaew, Co-Principal Investigator, University of Phayao
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: WP-5102031
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: Volunteer
MeSH Terms: interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aromatherapy (Experimental): Experimental procedures were conducted in the morning. Subjects individually entered the closed room where the temperature was kept at 25-26 oC and humidity 50-60%. The subjects were blinded using mask and were seated comfortably with eyes closed during experimental period. The EEG was recorded using silver electrodes. EEG activity was monitored 4 areas (F7, F8, T3 and T4) and ground electrodes. The experiments were divided into 3 parts. The first part, no-odor were recorded EEG activity for 10 minutes as a baseline. The second part, subject was exposure to the odor for 10 minutes as during inhalation. The last part, the odor was dispersed and assessed EEG activity for 10 minutes as after inhalation.
  Interventions: Other: Aromatherapy
- Pure water (Placebo Comparator): Experimental procedures were conducted in the morning. Subjects individually entered the closed room where the temperature was kept at 25-26 oC and humidity 50-60%. The subjects were blinded using mask and were seated comfortably with eyes closed during experimental period. The EEG was recorded using silver electrodes. EEG activity was monitored 4 areas (F7, F8, T3 and T4) and ground electrodes. The experiments were divided into 3 parts. The first part, no-odor were recorded EEG activity for 10 minutes as a baseline. The second part, subject was exposure to the water for 10 minutes as during inhalation. The last part, the water was dispersed and assessed EEG activity for 10 minutes as after inhalation.
  Interventions: Other: Pure water

INTERVENTIONS:
Other: Aromatherapy — Subject will assigned inhale aromatherapy
  Arms: Aromatherapy
Other: Pure water — Subject will assigned inhale Pure water
  Arms: Pure water

SUMMARY:
The purpose of this study is to examine and compare electroencephalography (EEG) changes in human subjects directly after inhalation of essential oils from five Thai aromatherapies. The investigators hypothesize that essential oils from Thai aromatherapies may influence the human EEG involving emotional relaxation particularly alpha wave EEG.

DETAILED DESCRIPTION:
The subjects consisted of 22 male and 26 female subjects , ages between 20 to 30 years (mean age, 23.3 years). They were screened for excessive nasal congestion, drug and food taken, and neurological disorders prior to participation in the experiment. The experiments were approved by the Ethical Committee for Research Involving Human Research Subject, Naresuan University. All subjects read and signed an informed consent before participation.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old

Exclusion Criteria:

* excessive nasal congestion
* neurological disorders prior to participation in the experiment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
electroencephalography (EEG) changes | baseline, 10 minutes
  The EEG was assessed for 10 minutes in each period; baseline, during and after inhaled the essential oil

CONTACTS AND LOCATIONS:
Overall Officials: Surasak Saokaew, PhD, Principal Investigator — University of Phayao
Locations (2):
- Thailand (2):
  - Surasak Saokaew, Muang, Changwat Phayao
  - University of Phayao, Muang, Changwat Phayao